CLINICAL TRIAL: NCT05791422
Title: Improvement of Low Back Pain After Surgical Decompression in Patients with Degenerative Lumbar Spinal Canal Stenosis
Brief Title: Improvement of Low Back Pain After Decompression in Patients with Degenerative Spinal Canal Stenosis
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Fayek Amin, Principle Investigator, Assiut University
Other Study IDs: LBPSD
Record Dates: First submitted 2023-03-15; First posted 2023-03-30 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2023-03

CONDITIONS: Low Back Pain; Lumbar Spinal Stenosis
MeSH Terms: conditions — Low Back Pain; Spinal Stenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Degenerative lumbar spine disease is a leading cause of disability in the world; it encompasses conditions such as spondylolisthesis, disc degeneration, and lumbar spinal stenosis. Those conditions present with a variety of clinical symptoms, including lower extremity pain, weakness, and low back pain (LBP) of varying levels of severity and in severe cases urine and stool incontinence may result.

DETAILED DESCRIPTION:
Degenerative lumbar spine disease is a common indication for lumbar decompression surgery, especially in elderly patients. Moreover, Clinical studies prove that decompression is superior to conservative treatment with more favorable outcomes .

Surgical options for decompressing the lumbar spine vary from minimally invasive disc decompression to open laminectomy and foraminotomy.

The surgery aims to improve the quality of life in appropriately selected patients , in the form of improvement of walking distance, lower limbs pain, and other symptoms of spinal compression.

Few papers assessed LBP improvement after lumbar decompression surgery . The common practice that patients with degenerative canal stenosis and low back pain should undergo fusion surgery is not evidence based.

In this study the investigators aim to assess the improvement of clinical symptoms, especially low back pain and lower limbs pain in patients with degenerative lumbar spine disease after undergoing lumbar decompression surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with degenerative lumbar spine disease admitted to Assiut University Hospitals, Department of Orthopaedic and Trauma Surgery between March 2023 and March 2024, to whom lumbar decompression surgery is indicated regardless of age or neurological symptoms.
2. Patients with grade one spondylolisthesis without evident instability can be added.

Exclusion Criteria:

1. Patients who are not available for follow up
2. Patients who refuse to participate in the study
3. Patients with evidence of instability
4. Previously operated patients on the same or adjacent segment.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with degenerative lumbar spine disease admitted to Assiut University Hospitals, Department of Orthopaedic and Trauma Surgery to whom lumbar decompression surgery is indicated .
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Changes in VAS score for low back pain following decompression surgery and in the follow up visits . | 1 year post operative
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

SECONDARY OUTCOMES:
Changes in ODI following decompression surgery and in the follow up visits. | 1 year post operative
  ODI is a 10-item self-assessing questionnaire, each item contains 6 levels of answers that can be scored from 0 to 5
Changes in EQ 5D 5l following decompression surgery and in the follow up visits. | 1 year post operative
  EQ-5D-5L is a descriptive system that comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit university hospitals, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Amundsen T, Weber H, Nordal HJ, Magnaes B, Abdelnoor M, Lilleas F. Lumbar spinal stenosis: conservative or surgical management?: A prospective 10-year study. Spine (Phila Pa 1976). 2000 Jun 1;25(11):1424-35; discussion 1435-6. doi: 10.1097/00007632-200006010-00016. PMID 10828926
- [Background] Berthelot JM, Bertrand-Vasseur A, Rodet D, Maugars Y, Prost A. Lumbar spinal stenosis: a review. Rev Rhum Engl Ed. 1997 May;64(5):315-25. PMID 9190005
- [Background] Arnoldi CC, Brodsky AE, Cauchoix J, Crock HV, Dommisse GF, Edgar MA, Gargano FP, Jacobson RE, Kirkaldy-Willis WH, Kurihara A, Langenskiold A, Macnab I, McIvor GW, Newman PH, Paine KW, Russin LA, Sheldon J, Tile M, Urist MR, Wilson WE, Wiltse LL. Lumbar spinal stenosis and nerve root entrapment syndromes. Definition and classification. Clin Orthop Relat Res. 1976 Mar-Apr;(115):4-5. No abstract available. PMID 1253495
- [Background] Athiviraham A, Yen D. Is spinal stenosis better treated surgically or nonsurgically? Clin Orthop Relat Res. 2007 May;458:90-3. doi: 10.1097/BLO.0b013e31803799a9. PMID 17308483
- [Background] Benz RJ, Garfin SR. Current techniques of decompression of the lumbar spine. Clin Orthop Relat Res. 2001 Mar;(384):75-81. doi: 10.1097/00003086-200103000-00010. PMID 11249182
- [Background] Sunderland G, Foster M, Dheerendra S, Pillay R. Patient-Reported Outcomes Following Lumbar Decompression Surgery: A Review of 2699 Cases. Global Spine J. 2021 Mar;11(2):172-179. doi: 10.1177/2192568219896541. Epub 2020 Jan 7. PMID 32875849
- [Background] Radcliff KE, Rihn J, Hilibrand A, DiIorio T, Tosteson T, Lurie JD, Zhao W, Vaccaro AR, Albert TJ, Weinstein JN. Does the duration of symptoms in patients with spinal stenosis and degenerative spondylolisthesis affect outcomes?: analysis of the Spine Outcomes Research Trial. Spine (Phila Pa 1976). 2011 Dec 1;36(25):2197-210. doi: 10.1097/BRS.0b013e3182341edf. PMID 21912308
- [Background] Jones AD, Wafai AM, Easterbrook AL. Improvement in low back pain following spinal decompression: observational study of 119 patients. Eur Spine J. 2014 Jan;23(1):135-41. doi: 10.1007/s00586-013-2964-5. Epub 2013 Aug 21. PMID 23963487
- [Background] Boonstra AM, Schiphorst Preuper HR, Reneman MF, Posthumus JB, Stewart RE. Reliability and validity of the visual analogue scale for disability in patients with chronic musculoskeletal pain. Int J Rehabil Res. 2008 Jun;31(2):165-9. doi: 10.1097/MRR.0b013e3282fc0f93. PMID 18467932
- [Background] Aburuz S, Bulatova N, Twalbeh M, Gazawi M. The validity and reliability of the Arabic version of the EQ-5D: a study from Jordan. Ann Saudi Med. 2009 Jul-Aug;29(4):304-8. doi: 10.4103/0256-4947.55313. PMID 19584581